CLINICAL TRIAL: NCT03750929
Title: Aerobic Capacity and Strength Exercise in Takayasu's Arteritis: Impact on Clinical, Laboratory and Vascular Parameters
Brief Title: Aerobic Capacity and Strength Exercise in Takayasu's Arteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Professor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MYO-HCFMUSP-05
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Physical Activity; Takayasu Arteritis
Keywords: Takayasus's arteritis; Physical exercises; Rheumatic diseases; Systemic vasculitis
MeSH Terms: conditions — Motor Activity; Takayasu Arteritis; Rheumatic Diseases; Systemic Vasculitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non physical exercises (No Intervention): Patients will not be submmitted to combined acute physical exercises (strength and aerobic)
- Physical exercises (Experimental): Patients will be submmitted to combined acute physical exercises (strength and aerobic) that consist on: supine, paddling, leg press 45º, knee extensor, flexor knee (two sets of 15 to 20 repetitions, with loads between 30% and 40% of a maximum repetition, with 30 seconds of interval). We will perform in the first exercise for upper and lower limbs, for heating, after starting the training where 4 series of 8 to 12 maximum repetitions will be performed, using the load between 70% and 80% of 1 maximum repetitions, already evaluated. The recovery between sets will be 90 seconds and between exercises will be 120 seconds.
  Interventions: Other: Combined acute physical exercises (strength and aerobic)

INTERVENTIONS:
Other: Combined acute physical exercises (strength and aerobic) — Patients will be submmitted to combined acute physical exercises (strength and aerobic)
  Arms: Physical exercises

SUMMARY:
Takayasu's arteritis is a primary systemic vasculitis that affects large vessels and their main branches. The objectives of the present study were to assess: a) the aerobic capacity (CA); b) security of the acute strength exercise session; c) correlation between CA, as well as strength exercise session, with demographic, clinical, therapeutic, comorbid parameters, and presence and degree of vascular damage; d) serum levels of the cytokines

DETAILED DESCRIPTION:
Takayasu's arteritis (TA) is a primary systemic vasculitis that affects large vessels and their main branches. It mainly affects young women. Blood vessel inflammation may result in stenosis, occlusions, ectasias and/or aneurysms and, consequently, difference of blood pressure between limbs and vascular claudication. Aerobic capacity (CA) is the measure of oxygen uptake, transport and use by the body, characterizing the individual's ability to perform activity. It is also a tool that can predict cardiovascular diseases. Our group has been a pioneer in demonstrating that CA is decreased in the small sample of the young women with TA. In addition, the safety and efficacy of aerobic exercises in this sample of patients were shown, as well as the influence of these sessions on the pro-inflammatory and angiogenic serum levels of the cytokines. However, due to the small samples, it was not possible to correlate CA with clinical and laboratory parameters and also with the presence of vascular damage. Moreover, to date, no studies have evaluated securityof an acute strength exercise session in TA.Therefore, thes objectives of the present study were to evaluate: a) the CA; b) security of the acute strength exercise session; c) correlation between CA, as well as strength exercise session, with demographic, clinical, therapeutic, comorbid parameters, and presence and degree of vascular damage; d) serum levels of the cytokine.

ELIGIBILITY:
Inclusion Criteria:

* Classification criteria of Takayasu's arteritis
* Sedentarism

Exclusion Criteria:

* Peripherical arterial diseases
* Non-controlled cardiovascular diseases
* Neurological diseases
* Patients with walking problem

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 12 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Security of acute session of combined physical exercises | One week before the exercises
  Acute aerobic with strength muscle test exercise

SECONDARY OUTCOMES:
Healthy Assessment Questionnaire (HAQ) | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  Especific questionnaire to assess the quality of life. Pontuaction: 0.00 (best) - 3.00 (worst).
Laboratory analysis (Serum levels of the protein C-reactive) | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  Protein C-reactive (< 5 mg/dL or not) will be analyzed to evaluate degree of disease activity
Indian Takayasu's Arteritis Activity Score (ITAS 2010) | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  Analyzing TA disease activity. Questionnaire with 44 items with 33 features arising from the cardiovascular system. Seven key items are weighted to score 2 and all others score 1 only. Activity was defined as ITAS 2010 score of ≥ 2 YES items
Cardiopulmonary test | Once (within 1 week before acute combined physical exercises)
  Patients will undertake a maximal graded exercise test on a treadmill, with increments in velocity and grade at every minute until volitional exhaustion (VO2) (mL/kg/minutes). VO2peak will be considered as the average of the final 30 seconds of the test.
Laboratory analysis (Erythrocyte rate sedimentation) | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  Erythrocyte rate sedimentation (reference: < 20 mm/ first hour) will be analyzed to evaluate degree of disease activity
Strength muscle tests 1 | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  The dynamic 1 maximum repetition for the bench-press exercises. The value of maximum repetition depending on each patient (unit: Newton).
Strength muscle tests 2 | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  The dynamic 1 maximum repetition for the leg-press press exercises. The value of maximum repetition depending on each patient (unit: Newton).
Strength muscle tests 3 | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  The dynamic 1 maximum repetition for the arm curl (with the dominant arm). The value of maximum repetition depending on each patient (unit: Newton).
Strength muscle tests 4 | Twice (within 1 week before and until 30 minutes after acute combined physical exercises)
  Isometric strength (assessed by handgrip, with the dominant arm) will be assessed. The value of maximum strenght will depend on each patient (unit: Newton).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel Katsuyuki Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided